CLINICAL TRIAL: NCT02850250
Title: Pharmacokinetics of Post Operative Cefuroxime in Infants Undergoing Cardiac Surgery
Acronym: PHOXEY
Status: Withdrawn | Type: Observational
Why Stopped: CI left the country so study has never opened
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PHOXEY
Record Dates: First submitted 2016-07-25; First posted 2016-07-29 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Event
Keywords: Observational; pharmacokinetic; cardiac; Cefuroxime; Paediatric
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cefuroxime; cefuroxime axetil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling on admission to PICU - then at 1 hour pre and post cefuroxime for 3 doses (8 hours apart)
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cefuroxime — Patients selected and treated as per normal pathway of care. Drugs will be prescribed as per standard Alder Hey Policy at the doses defined in the hospital policy Cefuroxime 50mg/kg 8 hourly (12 hourly if less than 7 days of age, or undergoing peritoneal dialysis - maximum 1.5grams per dose)
  Other Names: Ceftin

SUMMARY:
* To evaluate plasma concentrations of Cefuroxime in this patient population
* To determine if certain pathophysiological and/or iatrogenic conditions alter the pharmacokinetics in this patient group.
* To develop a rational physiological population pharmacokinetic model that describes plasma concentrations of medications in these patients.

DETAILED DESCRIPTION:
Congenital heart defects are structural or functional anomalies in the heart that occur during fetal development and are present at birth. Congenital heart disease is the most common congenital structural malformation. The survival of children born with congenital heart disease has improved dramatically over the past thirty years, improvements in diagnosis, medical and surgical management as well as anaesthetic care has improved survival rates from 20% to 80%.

Paediatric cardiac surgery Children with congenital heart disease may undergo either closed or open heart surgery. In a closed operation, the heart and main blood vessels can be operated on while the heart is still beating. In open procedures, the heart is opened and the blood flow to the child's vital organs is supported by a heart-lung bypass machine (Cardio-pulmonary bypass - CBP). In light of improving outcomes recent years has seen a worldwide shift towards neonatal biventricular repair where possible. For those where repair is not possible then the majority will be offered surgical univentricular palliation typically requiring 'high-risk' surgery in the first few weeks. 'High risk' neonates undergoing cardiac surgery often spend prolonged periods on the intensive care requiring maximal support.

These patients on the intensive care unit can suffer from multi-organ failure due to a variety of reasons and may require cardiovascular and respiratory support, and also renal replacement therapy in the form of peritoneal dialysis or haemodialysis/filtration. As a result of organ failure/support and different cardiac anatomy and physiology, the pharmacokinetics of drugs used in this post-operative period could potentially vary greatly.

Post-operative surgical site infections Post operative wound infections in paediatric patients undergoing cardiothoracic surgery occurs in 2.3% to 8% of patients. This complication results in increased morbidity, longer hospitalisations and increased cost. A major strategy in reducing postoperative surgical site infections has been the use of perioperative antibiotics to reduce primarily gram-positive skin flora that colonises the skin and can potentially infect an open wound.

Of particular concern for patients undergoing cardiac surgery are deep sternal wound infections or mediastinitis. Associated mortality is significant and has been reported to be as high as 60% in adults although there is little comparable data for children.

Neonates are at high risk of post-operative sternal wound infection, with an incidence of 5.5% versus 0.5% in older children in one study, which also highlighted an increased morbidity and mortality in the neonatal group.

Audit and data from our own institution has clarified that children aged less than 3 months at the time of surgery are at highest risk of developing a post-operative surgical site infection, and that the most commonly isolated organism is Staphylococcus Aureus.

Cefuroxime is the preferred choice of antibiotic prophylaxis in Alder Hey Children's Hospital. It is given intra-operatively, and post operatively for 24hours post, unless the patient's chest remains open, in which case the cefuroxime is continued until the chest is closed, or they are changed to another anti-microbial.

Pharmacokinetics of drugs in paediatric patients undergoing cardiac surgery Pharmacokinetics is a discipline aimed at predicting the best dosage and dosing regimen for each single drug in order to ensure and maintain therapeutically effective concentrations at the action sites.

In postoperative cardiac patients in critical care, there are a number of pathophysiological and iatrogenic conditions that may significantly alter the pharmacokinetic behavior of drugs.

These include -

* age
* weight
* temperature (if the patient is being actively cooled)
* single/biventricular circulations
* acute kidney injury
* passive peritoneal drainage
* active peritoneal dialysis
* continuous veno-venous haemofiltration/dialysis
* extra-corporeal membrane oxygenation

There is research available that paediatric patients undergoing cardiac surgery with cardio-pulmonary bypass (CPB) may have sub-therapeutic cefuroxime levels and the dose of cefuroxime should be adjusted accordingly.

In post op paediatric cardiac patients there are a number of studies describing different drug pharmacokinetics:

Dexmedetomidine pharmacokinetics may be influenced by age within the neonatal period, weight, total bypass time, and presence of intracardiac shunt.

Lower bodyweight was associated with lower epinephrine clearance. Milrinone clearance also appears to increase with age. Phenobarbital pharmacokinetics is also influenced by age and weight. Subjects with single ventricle physiology demonstrated a 15% decrease in clearance when compared with subjects with two-ventricle physiology.

So far to date, there are no pharmacokinetic studies investigating cefuroxime in this specific post-operative patient population.

Moreover, variations in the extracellular fluid content as a response to the trauma of surgery and the fluid load or significant drug loss through thoracic drainages or through PD catheter may significantly lower plasma concentrations of extracellularly distributed hydrophilic antimicrobials (beta-lactams, aminoglycosides and glycopeptides). Instability of renal function may promote significant changes in body fluid concentrations of renally eliminated drugs, even in a brief period of hours.

These factors cumulatively may lead to reduced or increased exposure to drugs. Dosages of some medicines are generally reduced in paediatric population following cardiac surgery to account for potential AKI (e.g. prophylactic antimicrobials), however potential losses through PD dialysis or through free drainage via PD catheter are not usually considered.

Passive Peritoneal Drainage/Peritoneal dialysis following paediatric cardiac surgery Children undergoing surgery for congenital heart disease are especially prone to acute kidney injury (AKI). It is difficult to appreciate the true incidence of this complication because, throughout the literature available, great variability is seen in the criteria used for the diagnosis. The reported incidence ranges between 1% and 17%, depending largely on the criteria used to define the condition, and the associated mortality is between 21% and 70%.

Peritoneal dialysis is commonly used in the post-operative period after cardiac surgery to aid the removal of fluids or sometimes as a treatment modality for acute kidney injury.

It is routine clinical practice in many centers, including ours (Department of Cardiac Surgery at Alder Hey Children's Hospital) to insert a peritoneal dialysis catheter electively at the time of surgery for potential peritoneal dialysis in neonates and children undergoing bypass surgery deemed to be at significant risk of needing post-operative PD. Following elective insertion of a PD catheter, hourly fluid drainage is documented as part of the routine ICU fluid balance charts. The vast majority will drain some fluid from the catheter in the initial hours. AKI usually develops early and PD is usually prescribed in the first days after the operation.

Between January 2014 until March 2015, 420 children underwent cardiac surgery at Alder Hey children's Hospital. Of these patients, 4% required PD in the post-operative period.

ECMO Occasionally patients are unable to be weaned from cardiopulmonary bypass following surgery, or deteriorate after arrival to intensive care and require Extracorporeal Membrane Oxygenation (ECMO). This group of patients have an increased volume of distribution and therefore, altered pharmacokinetic changes.

ELIGIBILITY:
Inclusion Criteria:

* Age from birth (>37 weeks gestation) to < 3 months
* Patients scheduled for congenital cardiac surgery and require cardiopulmonary bypass and intensive care admission post operatively in Alder Hey Children's Hospital
* Prescription of studied medications as per standard hospital policy.
* Intra-arterial catheter suitable for study sampling in situ.
* Informed consent by the parent or a legally authorised representative to participate in the study and to store specimens for immediate and future analysis.

Exclusion Criteria:

* No written informed consent
* Investigator's concerns
* Non English speaking
* No intra-arterial catheter

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged from birth (>37 weeks gestation) to < 3 months. Patients scheduled for congenital cardiac surgery and require cardiopulmonary bypass and intensive care admission post operatively in Alder Hey Children's Hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations | 12 months
  To measure plasma concentrations of Cefuroxime in this patient population

IPD SHARING:
Plan to Share IPD: Undecided
Undecided as yet